CLINICAL TRIAL: NCT03920852
Title: A Maximum Use Trial of Ruxolitinib Cream in Adolescent and Adult Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-103
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; ruxolitinib cream; maximum use
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib cream (Experimental)
  Interventions: Drug: Ruxolitinib cream

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib 1.5% cream applied twice daily.
  Other Names: INCB018424 phosphate cream

SUMMARY:
This is an open-label maximum use trial to evaluate ruxolitinib safety and blood levels after its topical application twice daily to affected areas (≥ 25% BSA) in adolescent and adult participants with atopic dermatitis (AD) and to determine if its systemic bioavailability results in any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with atopic dermatitis as defined by Hanifin and Rajka criteria.
* Atopic dermatitis duration of at least 2 years.
* Investigator's Global Assessment score of at least 2 at screening and baseline.
* Body surface area of atopic dermatitis involvement of ≥ 25% at screening and baseline.
* Agree to discontinue all agents used to treat atopic dermatitis from screening through the final follow up visit.
* Willing to take appropriate contraceptive measures to avoid pregnancy or fathering a child for the duration of study participation with the exception of females of nonchildbearing potential and prepubescent adolescents.
* Written informed consent of the participant or parent(s)/legal guardian and a verbal or written assent from the participant when possible.

Exclusion Criteria:

* Unstable course of atopic dermatitis (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks before baseline.
* Concurrent conditions and history of other diseases:

  * Immunocompromised (eg, lymphoma, acquired immunodeficiency syndrome, Wiskott-Aldrich syndrome).
  * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 14 days (2 weeks) before the baseline visit.
  * Active acute bacterial, fungal, or viral (eg, herpes simplex, herpes zoster, chicken pox) skin infection within 7 days (1 week) before the baseline visit.
  * Any other concomitant skin disorder (eg, generalized erythroderma, such as Netherton syndrome, or psoriasis), pigmentation, or extensive scarring that in the opinion of the investigator may interfere with the evaluation of AD lesions or compromise participant safety.
  * Other types of eczema.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full study participation, pose a significant risk to the participant, or interfere with interpretation of study data.
* Use of any of the following treatments within the indicated washout periods before baseline:

  * 5 half-lives or 84 days (12 weeks), whichever is longer: biologic agents (eg, dupilumab).
  * 28 days (4 weeks): systemic corticosteroids or adrenocorticotropic hormone analogues, cyclosporine, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (eg, mycophenolate or tacrolimus).
  * 14 days (2 weeks) or 5 half-lives, whichever is longer: immunizations and sedating antihistamines, unless on long-term stable regimen (nonsedating antihistamines are permitted); and potent systemic CYP3A4 inhibitors or fluconazole.
  * 7 days (1 week): other topical treatments applied onto atopic dermatitis skin lesions (other than bland emollients), such as corticosteroids, crisaborole, calcineurin inhibitors, coal tar (shampoo), antibiotics, antibacterial cleansing body wash/soap.
* Treatment with Janus kinase inhibitors (systemic or topical) within 12 weeks (3 months) from baseline.
* Ultraviolet light therapy or prolonged exposure to natural or artificial sources of ultraviolet radiation (eg, sunlight or tanning booth) within 14 days (2 weeks) before baseline and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the participant's atopic dermatitis.
* Positive serology test results at screening for HIV antibody.
* Liver function test results outside the protocol-defined range.
* Pregnant or lactating participants or those considering pregnancy.
* History of alcoholism or drug addiction within 365 days (1 year) before screening or current alcohol or drug use that, in the opinion of the investigator, will interfere with the participant's ability to comply with the administration schedule and study assessments.
* Current treatment or treatment within 28 days (4 weeks) or 5 half-lives (whichever is longer) before the baseline visit with another investigational medication or current enrollment in another investigational drug protocol.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Up to 127 days
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first application of study drug.

SECONDARY OUTCOMES:
Plasma concentration of ruxolitinib | Up to 127 days
Cmax of ruxolitinib | Up to 127 days
  Maximum measured plasma concentration.
Tmax of ruxolitinib | Up to 127 days
  Time to achieve the observed maximum plasma concentration.
AUC0-12 of ruxolitinib | Up to 127 days
  Area under the concentration-time curve from 0 to 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Kuligowski, MD, Study Director — Incyte Corporation
Locations (10):
- United States (9):
  - Orange County Research Center, Anaheim, California
  - Encino Research Center, Encino, California
  - RM Medical Research, INC., Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Pure Skin Dermatology Aesthetics at Accel Research, Orlando, Florida
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Oakland Hills Dermatology PC, Auburn Hills, Michigan
  - Clinical Research Institute of Southern Oregon - Crisor, Medford, Oregon
  - Clinical Research Partners LLC, Richmond, Virginia
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bissonnette R, Call RS, Raoof T, Zhu Z, Yeleswaram S, Gong X, Lee M. A Maximum-Use Trial of Ruxolitinib Cream in Adolescents and Adults with Atopic Dermatitis. Am J Clin Dermatol. 2022 May;23(3):355-364. doi: 10.1007/s40257-022-00690-3. Epub 2022 Apr 4. PMID 35368221
- [Derived] Scuron MD, Fay BL, Connell AJ, Peel MT, Smith PA. Ruxolitinib Cream Has Dual Efficacy on Pruritus and Inflammation in Experimental Dermatitis. Front Immunol. 2021 Feb 15;11:620098. doi: 10.3389/fimmu.2020.620098. eCollection 2020. PMID 33658996